CLINICAL TRIAL: NCT00944229
Title: Salutary Effects of Dietary Supplementation With OMEGA 3 on Exercise Performance and Endothelial Function in Patients With Congestive Heart Failure. A Matter of Lipid Oxidation ?
Brief Title: The Effect of Omega-3 Polyunsaturated Fatty Acids in Congestive Heart Failure
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: PI left the institution
Sponsor: Columbia University (Other)
Collaborators: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: AAAD7501; LVZ112854 (Other: GSK protocol #)
Record Dates: First submitted 2009-02-12; First posted 2009-07-23 (Estimated); Results first posted 2016-04-22 (Estimated); Last update posted 2016-05-25 (Estimated); Status verified 2016-04

CONDITIONS: Heart Failure
Keywords: Heart Failure; omega 3; lovaza; VO2 max
MeSH Terms: conditions — Heart Failure | interventions — Omacor; Docosahexaenoic Acids

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 Drug Treatment - LOVAZA (Active Comparator): Drug Treatment - LOVAZA 4 gm q24 for 8 weeks
  Interventions: Drug: LOVAZA (Omega-3)
- 2 placebo (Placebo Comparator): Placebo 4 capsules q24 for 8 weeks
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: LOVAZA (Omega-3) — LOVAZA 4 gm q24 for 8 weeks Each 1-gram capsule of LOVAZA (omega-3-acid ethyl esters) contains at least 900 mg of the ethyl esters of omega-3 fatty acids. These are predominantly a combination of ethyl esters of eicosapentaenoic acid (EPA - approximately 465 mg) and docosahexaenoic acid (DHA - approximately 375 mg).
  Arms: 1 Drug Treatment - LOVAZA
Drug: Placebo — 4 capsules of placebo every 24 hours
  Arms: 2 placebo

SUMMARY:
A diet rich in Omega-3 (fish oil) reduces plasma triglycerides and the risk for ischemic heart disease. Recently, a large trial evaluating treatment with Omega 3 in heart failure patients suggested that omega 3 may lower the risk of death from CHF. The mechanism of this potential benefit is not well understood.

Methods:

Forty patients will be enrolled in the study. Twenty patients will receive Omega 3 (lovaza 4 gm a day) and 20 patients will receive placebo. All subjects will have assessment of their exercise capacity and blood vessel function before and after an 8 week treatment period. About 4 table spoons of blood will be drawn throughout the study.

Expected results:

The investigators believe that omega 3 may improve the ability to exercise and improve blood vessel function.

DETAILED DESCRIPTION:
A diet rich in Omega-3 polyunsaturated fatty acids Omega 3 reduces plasma triglycerides and the risk for ischemic heart disease1, and may exert direct antiarrhythmic effect on the myocardium 2-9. A post-hoc analysis of the GISSI-Prevenzione trial demonstrated a reduction in all-cause and sudden mortality in a subgroup of nearly 2000 post-infarction patients with left ventricular dysfunction 10. This provocative finding has now been prospectively studied in a large-scale, randomized, double-blind study designed to investigate the effects of Omega 3 on mortality and morbidity in patients with symptomatic heart failure (the GISSI Heart Failure project). The results of the GISSI-HF trial demonstrate that 1 g per day of Omega 3 is associated with 9% reduction in mortality and cardiovascular admissions in patients with predominantly systolic heart failure, when added to optimal medical therapy11.

The mechanism(s) underlying these beneficial effects remains to be elucidated and will be critical in fully exhausting the therapeutic benefits of Omega 3 in CHF. We have recently demonstrated that lipid oxidation during acute exercise is altered in patients with CHF 12 and that the degree of this alteration carries prognostic significance. It is conceivable that Omega 3 modulates lipid oxidation during exercise and thereby favorably effect outcome. Accordingly we propose to study the effect of Omega 3 on lipid oxidation during exercise in CHF. We will further examine VO2 and endothelial function at present the principal surrogate markers for survival in CHF 13.

ELIGIBILITY:
Inclusion Criteria:

All subjects with CHF due to systolic dysfunction followed at the outpatient facilities of Columbia University Medical Center will be screened and subjects will be asked to participate if the following criteria are met:

* Older than 18 years.
* Symptomatic heart failure (New York Heart Association functional class II-III).
* Ischemic or non-ischemic cardiomyopathy.
* Left ventricular ejection fraction (EF) 40% or lower.
* Peak oxygen uptake (VO2, peak) between 10 and 17 mL O2/min/kg.
* Be on appropriate, stable medical treatments for heart failure, including (unless shown to be intolerant) a diuretic, an angiotensin-converting enzyme inhibitor and/or angiotensin-receptor blocker and a beta-blocker, pacemaker or ICD or CRT.

Exclusion Criteria:

* Unable to perform treadmill exercise
* Pregnancy
* Recent myocardial infarction (within 3 months).
* Clinically significant angina.
* Hospitalization for heart failure requiring intravenous treatments within 30 days.
* Allergy to fish

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 58 (Actual)
Dates: Start 2010-01; Primary Completion 2014-03 (Actual); Study Completion 2014-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ulrich Jorde, MD, Principal Investigator — Columbia University
Locations (1):
- Columbia University Medical Center, New York, New York, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The principal investigator has left the institution. Attempts to contact the PI have been unsuccessful. Columbia will never have access to the data. Thus, data will not be analyzed. The only information available is the number of participants who started and completed the study, which was last reported to and approved by the IRB in March 2013.
Groups:
- LOVAZA or Placebo: Data per arm is not available. Columbia will never have access to this data.
Period: Overall Study
Arm/Group | LOVAZA or Placebo
Started | 58
Completed | 33
Not Completed | 25
Not completed — Withdrawal by Subject | 11
Not completed — Physician Decision | 14

BASELINE CHARACTERISTICS:
Arm/Group | LOVAZA or Placebo
Number analyzed (Participants) | 58
Age, Customized [Number; unit: participants]
  Between 18 and 65 years | 50
  >=65 years | 8
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 22
  Male | 36
Race/Ethnicity, Customized [Number; unit: participants]
  African American | 13
  Asian | 3
  Caucasian | 28
  Hispanic | 14
Region of Enrollment [Number; unit: participants]
  United States | 58

OUTCOME MEASURES:

1. Primary Outcome: Change in Peak VO2
Time Frame: 0, 1 and 8 weeks of Omega 3 supplementation.
Population: The principal investigator has left the institution. Attempts to contact the PI have been unsuccessful. Columbia will never have access to the data. Thus, data will not be analyzed. The only information available is the number of participants who started and completed the study, which was last reported to and approved by the IRB in March 2013.
Arm/Group | LOVAZA or Placebo
Number analyzed (Participants) | 0

2. Primary Outcome: Change in Reactive Hyperemia Peripheral Arterial Tonometry (RH-PAT) After 8 Weeks of Omega 3 Supplementation.
Time Frame: 0 and after 8 weeks of Omega 3 supplementation.
Population: as for outcome 1
Arm/Group | LOVAZA or Placebo
Number analyzed (Participants) | 0

3. Primary Outcome: Change in Base Line Oxidized Low Density Lipoprotein (LDL) Level and in Response to Exercise
Time Frame: 0, 1 and 8 weeks of Omega 3 supplementation.
Population: as for outcome 1
Arm/Group | LOVAZA or Placebo
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Description: The principal investigator has left the institution. Attempts to contact the PI have been unsuccessful. Columbia will never have access to the data. Thus, data will not be analyzed. The only information available is the number of participants who started and completed the study, which was last reported to and approved by the IRB in March 2013.
Arm/Group | LOVAZA or Placebo
Serious Adverse Events (participants affected / at risk) | 0/0
Other Adverse Events (participants affected / at risk) | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No